CLINICAL TRIAL: NCT04379921
Title: Improving Spine Surgical Care With Real-Time Objective Patient Tracking Using the Apple Watch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Principal Investigator, Corinna Zygourakis, Assistant Professor of Neurosurgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 52367
Record Dates: First submitted 2020-04-30; First posted 2020-05-08 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-03

CONDITIONS: Spine Disease; Spine Degeneration; Spinal Stenosis; Surgery; Spine Fusion
Keywords: Spine Surgery; Apple Watch; Objective Tracking of Spine Surgery Outcomes
MeSH Terms: conditions — Spinal Diseases; Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): Participants will receive standard care.
- Apple Watch and App (Experimental): Participants will receive standard care, and an Apple Watch to record activity through the App.
  Interventions: Device: Apple Watch and App

INTERVENTIONS:
Device: Apple Watch and App — Participants in the Apple Watch and App arm will receive an Apple Watch and download an App (NeuroCoach). The Apple Watch and App are used for this study to record patient's mobility information (e.g., step counts, heart rate, stairs climbed, distance traveled) as well as provide an additional platform for patients to complete questionnaires.
  Arms: Apple Watch and App

SUMMARY:
One of the primary goals of spine surgery is to reduce pain and increase mobility to improve patients' quality of life. Currently, there is no established method for surgeons to objectively track their patients' mobilization postoperatively. This study is the first prospective trial utilizing the Apple Watch to objectively track patients before and after elective spine surgery. The investigators hypothesize that the ability of patients to track their own activity and discuss with their surgeon objective mobilization goals will not only help patients achieve empowerment in their own care but also improve their overall satisfaction and self-reported outcomes after spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking.
* Undergoing elective spine surgery by attending physicians at Stanford University.
* Own iPhone

Exclusion Criteria:

* Patients with spine trauma, tumors, or infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corinna Zygourakis, MD, Principal Investigator — Department of Neurosurgery at Stanford University
Locations (1):
- Stanford University Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernstein DN, Brodell D, Li Y, Rubery PT, Mesfin A. Impact of the Economic Downturn on Elective Lumbar Spine Surgery in the United States: A National Trend Analysis, 2003 to 2013. Global Spine J. 2017 May;7(3):213-219. doi: 10.1177/2192568217694151. Epub 2017 Apr 6. PMID 28660102
- [Background] Davis H. Increasing rates of cervical and lumbar spine surgery in the United States, 1979-1990. Spine (Phila Pa 1976). 1994 May 15;19(10):1117-23; discussion 1123-4. doi: 10.1097/00007632-199405001-00003. PMID 8059266
- [Background] O'Lynnger TM, Zuckerman SL, Morone PJ, Dewan MC, Vasquez-Castellanos RA, Cheng JS. Trends for Spine Surgery for the Elderly: Implications for Access to Healthcare in North America. Neurosurgery. 2015 Oct;77 Suppl 4:S136-41. doi: 10.1227/NEU.0000000000000945. PMID 26378351
- [Background] Parker SL, Chotai S, Devin CJ, Tetreault L, Mroz TE, Brodke DS, Fehlings MG, McGirt MJ. Bending the Cost Curve-Establishing Value in Spine Surgery. Neurosurgery. 2017 Mar 1;80(3S):S61-S69. doi: 10.1093/neuros/nyw081. PMID 28350948
- [Background] Epstein NE. A review article on the benefits of early mobilization following spinal surgery and other medical/surgical procedures. Surg Neurol Int. 2014 Apr 16;5(Suppl 3):S66-73. doi: 10.4103/2152-7806.130674. eCollection 2014. PMID 24843814
- [Background] Guzman JZ, Cutler HS, Connolly J, Skovrlj B, Mroz TE, Riew KD, Cho SK. Patient-Reported Outcome Instruments in Spine Surgery. Spine (Phila Pa 1976). 2016 Mar;41(5):429-37. doi: 10.1097/BRS.0000000000001211. PMID 26571179
- [Background] Lu TC, Fu CM, Ma MH, Fang CC, Turner AM. Healthcare Applications of Smart Watches. A Systematic Review. Appl Clin Inform. 2016 Sep 14;7(3):850-69. doi: 10.4338/ACI-2016-03-R-0042. PMID 27623763
- [Background] Reeder B, David A. Health at hand: A systematic review of smart watch uses for health and wellness. J Biomed Inform. 2016 Oct;63:269-276. doi: 10.1016/j.jbi.2016.09.001. Epub 2016 Sep 6. PMID 27612974
- [Background] Henriksen A, Haugen Mikalsen M, Woldaregay AZ, Muzny M, Hartvigsen G, Hopstock LA, Grimsgaard S. Using Fitness Trackers and Smartwatches to Measure Physical Activity in Research: Analysis of Consumer Wrist-Worn Wearables. J Med Internet Res. 2018 Mar 22;20(3):e110. doi: 10.2196/jmir.9157. PMID 29567635
- [Background] Mobbs RJ, Phan K, Maharaj M, Rao PJ. Physical Activity Measured with Accelerometer and Self-Rated Disability in Lumbar Spine Surgery: A Prospective Study. Global Spine J. 2016 Aug;6(5):459-64. doi: 10.1055/s-0035-1565259. Epub 2015 Oct 13. PMID 27433430
- [Background] Phan K, Mobbs RJ. Long-Term Objective Physical Activity Measurements using a Wireless Accelerometer Following Minimally Invasive Transforaminal Interbody Fusion Surgery. Asian Spine J. 2016 Apr;10(2):366-9. doi: 10.4184/asj.2016.10.2.366. Epub 2016 Apr 15. PMID 27114781
- [Background] Breteler MJ, Janssen JH, Spiering W, Kalkman CJ, van Solinge WW, Dohmen DA. Measuring Free-Living Physical Activity With Three Commercially Available Activity Monitors for Telemonitoring Purposes: Validation Study. JMIR Form Res. 2019 Apr 24;3(2):e11489. doi: 10.2196/11489. PMID 31017587
- [Background] Veerabhadrappa P, Moran MD, Renninger MD, Rhudy MB, Dreisbach SB, Gift KM. Tracking Steps on Apple Watch at Different Walking Speeds. J Gen Intern Med. 2018 Jun;33(6):795-796. doi: 10.1007/s11606-018-4332-y. PMID 29633143
- [Background] Xie J, Wen D, Liang L, Jia Y, Gao L, Lei J. Evaluating the Validity of Current Mainstream Wearable Devices in Fitness Tracking Under Various Physical Activities: Comparative Study. JMIR Mhealth Uhealth. 2018 Apr 12;6(4):e94. doi: 10.2196/mhealth.9754. PMID 29650506
- [Derived] Maldaner N, Tang M, Fatemi P, Leung C, Desai A, Tomkins-Lane C, Zygourakis C. Standardizing Physical Activity Monitoring in Patients With Degenerative Lumbar Disorders. Neurosurgery. 2024 Apr 1;94(4):788-796. doi: 10.1227/neu.0000000000002755. Epub 2023 Nov 13. PMID 37955445
- See also: 2017 Profile of Older Americans — https://acl.gov/sites/default/files/Aging%20and%20Disability%20in%20America/2017OlderAmericansProfile.pdf
- See also: Global Smartwatch Vendor Market Share — https://www.strategyanalytics.com/access-services/devices/wearables/market-data/report-detail/global-smartwatch-vendor-market-share-by-region-q4-2018

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Participants receive standard care.
- Apple Watch and App: Participants receive standard care, and an Apple Watch to record activity through the NeuroCoach App, recording patient's mobility information (e.g., step counts, heart rate, stairs climbed, distance traveled) as well as provide an additional platform for patients to complete questionnaires.
Period: Overall Study
Arm/Group | Control | Apple Watch and App
Started | 122 | 133
Completed | 96 | 96
Not Completed | 26 | 37

BASELINE CHARACTERISTICS:
Population: Participants who completed 12 month assessments
Groups:
- Apple Watch and App: Participants receive standard care, and an Apple Watch to record activity through the NeuroCoach App.
- Total: Total of all reporting groups
Arm/Group | Control | Apple Watch and App | Total
Number analyzed (Participants) | 91 | 96 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.03 (13.22) | 61.79 (13.28) | 60.46 (13.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 58 | 108
  Male | 41 | 38 | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Self-reported by patient
  Participants
    Asian | 7 | 6 | 13
    Black or African American | 1 | 5 | 6
    Hispanic and Asian | 2 | 0 | 2
    Hispanic and Latino | 5 | 7 | 12
    Native Hawaiians and Other Pacific Islanders | 0 | 1 | 1
    Other | 7 | 8 | 15
    Unknown | 0 | 0 | 0
    White | 67 | 67 | 134
    White and Hispanic | 2 | 1 | 3
    White and Native American | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 91 | 96 | 187

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Objective Patient Measures (Steps, Distance Travelled, From Apple Watch) and Patient-Reported Outcome Measures (SF-36, EQ-5D, PROMIS, NDI, ODI)
Description: Steps and distance (meters) collected by Apple Watch were averaged across the outcome measure time frame. Survey scores were collected at the end of the outcome measure time frame.
  * Short Form-36 (SF-36): Scores range from 0 to 100. Higher scores indicate better health outcomes.
  * EuroQOL-5 Dimensional Questionnaire (EQ-5D): Scores range from 0 to 100. Higher scores indicate better health outcomes.
  * Patient-Reported Outcomes Measurement Information System (PROMIS): Scores range from 41 to 78.3. Higher scores indicate worse health outcomes.
  * Neck Disability Index (NDI): Scores range from 0 to 100. Higher scores indicate worse health outcomes.
  * Oswestry Disability Index (ODI): Scores range from 0 to 100. Higher scores indicate worse health outcomes.
Time Frame: 2-6 weeks pre-operatively
Population: Participants with data for the respective time frame and patient-reported outcome. This outcome was evaluated on the Apple Watch and App group only (the Control group was not assigned an Apple Watch).
Measure: Number; unit: correlation coefficient
Arm/Group | Apple Watch and App
Number analyzed (Participants) | 90
correlation coefficient
  Steps to SF-36 | 0.160804476
  Steps to EQ-5D | 0.170547163
  Steps to PROMIS | 0.03133065
  Steps to NDI: number analyzed (Participants) | 30
  Steps to NDI | -0.287227624
  Steps to ODI: number analyzed (Participants) | 53
  Steps to ODI | -0.245495419
  Distance traveled (meters) to SF-36 | 0.156072138
  Distance traveled (meters) to EQ-5D | 0.165543596
  Distance traveled (meters) to PROMIS | 0.047067760
  Distance traveled (meters) to NDI: number analyzed (Participants) | 30
  Distance traveled (meters) to NDI | -0.288155169
  Distance traveled (meters) to ODI: number analyzed (Participants) | 53
  Distance traveled (meters) to ODI | -0.238599412
Statistical Analysis 1: Comparison: Apple Watch and App; Analysis of correlation: steps to SF-36; Test type: Other; p = 0.26801155, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is < 0.05. The p-value is adjusted using the Benjamini-Hochberg (BH method)
Statistical Analysis 2: Comparison: Apple Watch and App; Analysis of correlation: steps to EQ-5D; Test type: Other; p = 0.27520264, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Apple Watch and App; Analysis of correlation: steps to PROMIS; Test type: Other; p = 0.95547874, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Apple Watch and App; Analysis of correlation: steps to NDI; Test type: Other; p = 0.56230120, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Apple Watch and App; Analysis of correlation: steps to ODI; Test type: Other; p = 0.35813970, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to SF-36; Test type: Other; p = 0.26801155, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to EQ-5D; Test type: Other; p = 0.08121447, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to PROMIS; Test type: Other; p = 0.95547874, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to NDI; Test type: Other; p = 0.59932922, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to ODI; Test type: Other; p = 0.35813970, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Correlation Between Objective Patient Measures (Steps, Distance Travelled, From Apple Watch) and Patient-Reported Outcome Measures (SF-36, EQ-5D, PROMIS, NDI, ODI)
Description: as for outcome 1
Time Frame: 4-6 weeks post-operatively
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Apple Watch and App
Number analyzed (Participants) | 88
correlation coefficient
  Steps to SF-36 | 0.237509597
  Steps to EQ-5D | 0.254596876
  Steps to PROMIS | -0.061318768
  Steps to NDI: number analyzed (Participants) | 29
  Steps to NDI | -0.026754947
  Steps to ODI: number analyzed (Participants) | 42
  Steps to ODI | -0.237678247
  Distance traveled (meters) to SF-36 | 0.251030049
  Distance traveled (meters) to EQ-5D | 0.249053662
  Distance traveled (meters) to PROMIS | -0.044081635
  Distance traveled (meters) to NDI: number analyzed (Participants) | 29
  Distance traveled (meters) to NDI | -0.047181840
  Distance traveled (meters) to ODI: number analyzed (Participants) | 42
  Distance traveled (meters) to ODI | -0.234325616
Statistical Analysis 1: Comparison: Apple Watch and App; Analysis of correlation: steps to SF-36; Test type: Other; p = 0.09091440, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Apple Watch and App; Analysis of correlation: steps to EQ-5D; Test type: Other; p = 0.12858419, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Apple Watch and App; Analysis of correlation: steps to PROMIS; Test type: Other; p = 0.95547874, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Apple Watch and App; Analysis of correlation: steps to NDI; Test type: Other; p = 0.93040170, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Apple Watch and App; Analysis of correlation: steps to ODI; Test type: Other; p = 0.38647114, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to SF-36; Test type: Other; p = 0.09091440, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to EQ-5D; Test type: Other; p = 0.12858419, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to PROMIS; Test type: Other; p = 0.95547874, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to NDI; Test type: Other; p = 0.93040170, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to ODI; Test type: Other; p = 0.38647114, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Correlation Between Objective Patient Measures (Steps, Distance Travelled, From Apple Watch) and Patient-Reported Outcome Measures (SF-36, EQ-5D, PROMIS, NDI, ODI)
Description: as for outcome 1
Time Frame: 6 weeks-3 months post-operatively
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Apple Watch and App
Number analyzed (Participants) | 85
correlation coefficient
  Steps to SF-36 | 0.211745206
  Steps to EQ-5D | 0.137757731
  Steps to PROMIS | -0.028651640
  Steps to NDI: number analyzed (Participants) | 29
  Steps to NDI | -0.195235044
  Steps to ODI: number analyzed (Participants) | 44
  Steps to ODI | -0.130278276
  Distance traveled (meters) to SF-36 | 0.205169697
  Distance traveled (meters) to EQ-5D | 0.122267044
  Distance traveled (meters) to PROMIS | -0.004087870
  Distance traveled (meters) to NDI: number analyzed (Participants) | 29
  Distance traveled (meters) to NDI | -0.195274715
  Distance traveled (meters) to ODI: number analyzed (Participants) | 44
  Distance traveled (meters) to ODI | -0.102500089
Statistical Analysis 1: Comparison: Apple Watch and App; Analysis of correlation: steps to SF-36; Test type: Other; p = 0.14778771, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Apple Watch and App; Analysis of correlation: steps to EQ-5D; Test type: Other; p = 0.36288455, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Apple Watch and App; Analysis of correlation: steps to PROMIS; Test type: Other; p = 0.95547874, Wilcoxon (Mann-Whitney); The a priori threshold for statistical significance is < 0.05. The p-value is adjusted using the Benjamini-Hochberg (BH method)
Statistical Analysis 4: Comparison: Apple Watch and App; Analysis of correlation: steps to NDI; Test type: Other; p = 0.65291937, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Apple Watch and App; Analysis of correlation: steps to ODI; Test type: Other; p = 0.61429132, Wilcoxon (Mann-Whitney); [statistical method as in outcome 3, analysis 3]
Statistical Analysis 6: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to SF-36; Test type: Other; p = 0.15896420, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to EQ-5D; Test type: Other; p = 0.39253325, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to PROMIS; Test type: Other; p = 0.99526258, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to NDI; Test type: Other; p = 0.65291937, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to ODI; Test type: Other; p = 0.67694276, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

4. Primary Outcome: Correlation Between Objective Patient Measures (Steps, Distance Travelled, From Apple Watch) and Patient-Reported Outcome Measures (SF-36, EQ-5D, PROMIS, NDI, ODI)
Description: as for outcome 1
Time Frame: 3-6 months post-operatively
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Apple Watch and App
Number analyzed (Participants) | 77
correlation coefficient
  Steps to SF-36 | 0.299619225
  Steps to EQ-5D | 0.313524073
  Steps to PROMIS | -0.086753507
  Steps to NDI: number analyzed (Participants) | 27
  Steps to NDI | -0.239505761
  Steps to ODI: number analyzed (Participants) | 35
  Steps to ODI | -0.322504210
  Distance traveled (meters) to SF-36 | 0.293769111
  Distance traveled (meters) to EQ-5D | 0.308525815
  Distance traveled (meters) to PROMIS | -0.067371364
  Distance traveled (meters) to NDI: number analyzed (Participants) | 27
  Distance traveled (meters) to NDI | -0.234173267
  Distance traveled (meters) to ODI: number analyzed (Participants) | 35
  Distance traveled (meters) to ODI | -0.325285216
Statistical Analysis 1: Comparison: Apple Watch and App; Analysis of correlation: steps to SF-36; Test type: Other; p = 0.06340316, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Apple Watch and App; Analysis of correlation: steps to EQ-5D; Test type: Other; p = 0.08121447, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Apple Watch and App; Analysis of correlation: steps to PROMIS; Test type: Other; p = 0.95547874, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Apple Watch and App; Analysis of correlation: steps to NDI; Test type: Other; p = 0.59932922, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Apple Watch and App; Analysis of correlation: steps to ODI; Test type: Other; p = 0.35813970, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to SF-36; Test type: Other; p = 0.06340316, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to EQ-5D; Test type: Other; p = 0.08121447, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to PROMIS; Test type: Other; p = 0.95547874, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to NDI; Test type: Other; p = 0.59932922, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to ODI; Test type: Other; p = 0.35813970, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

5. Primary Outcome: Correlation Between Objective Patient Measures (Steps, Distance Travelled, From Apple Watch) and Patient-Reported Outcome Measures (SF-36, EQ-5D, PROMIS, NDI, ODI)
Description: as for outcome 1
Time Frame: 6-12 months post-operatively
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Apple Watch and App
Number analyzed (Participants) | 73
correlation coefficient
  Steps to SF-36: number analyzed (Participants) | 72
  Steps to SF-36 | 0.093993286
  Steps to EQ-5D | 0.144224016
  Steps to PROMIS | -0.094520314
  Steps to NDI: number analyzed (Participants) | 26
  Steps to NDI | 0.055377523
  Steps to ODI: number analyzed (Participants) | 38
  Steps to ODI | -0.257180828
  Distance traveled (meters) to SF-36: number analyzed (Participants) | 72
  Distance traveled (meters) to SF-36 | 0.058395557
  Distance traveled (meters) to EQ-5D | 0.153422291
  Distance traveled (meters) to PROMIS | -0.109789378
  Distance traveled (meters) to NDI: number analyzed (Participants) | 26
  Distance traveled (meters) to NDI | 0.027880729
  Distance traveled (meters) to ODI: number analyzed (Participants) | 38
  Distance traveled (meters) to ODI | -0.202307765
Statistical Analysis 1: Comparison: Apple Watch and App; Analysis of correlation: steps to SF-36; Test type: Other; p = 0.52394318, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Apple Watch and App; Analysis of correlation: steps to EQ-5D; Test type: Other; p = 0.37244637, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Apple Watch and App; Analysis of correlation: steps to PROMIS; Test type: Other; p = 0.95547874, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Apple Watch and App; Analysis of correlation: steps to NDI; Test type: Other; p = 0.93040170, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Apple Watch and App; Analysis of correlation: steps to ODI; Test type: Other; p = 0.38647114, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to SF-36; Test type: Other; p = 0.71552390, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to EQ-5D; Test type: Other; p = 0.35456143, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to PROMIS; Test type: Other; p = 0.95547874, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to NDI; Test type: Other; p = 0.93040170, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Apple Watch and App; Analysis of correlation: distance (meters) to ODI; Test type: Other; p = 0.42512141, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

6. Primary Outcome: Change in Objective Outcome Measures: Number of Steps After Surgery
Description: Steps per day collected by Apple Watch were averaged across the respective outcome measure time frame. Change was calculated as the post-baseline value minus the baseline value (which was normalized to zero).
Time Frame: 2-6 weeks pre-operatively; 4-6 weeks, 6 weeks-3 months, 3-6 months, and 6-12 months post-operatively
Population: Participants with available data at the respective time point. This outcome was evaluated on the Apple Watch and App group only (the Control group was not assigned an Apple Watch).
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Apple Watch and App
Number analyzed (Participants) | 88
steps per day
  4-6 weeks post-operatively | -1166.04 (2272.07)
  6 weeks-3 months post-operatively: number analyzed (Participants) | 85
  6 weeks-3 months post-operatively | 764.68 (2066.11)
  3-6 months post-operatively: number analyzed (Participants) | 77
  3-6 months post-operatively | 1212.10 (2177.45)
  6-12 months post-operatively: number analyzed (Participants) | 73
  6-12 months post-operatively | 1068.73 (2048.83)

7. Primary Outcome: Change in Objective Outcome Measures: Distance Traveled (Meters) After Surgery
Description: Meters per day collected by Apple Watch were averaged across the respective outcome measure time frame. Change was calculated as the post-baseline value minus the baseline value (which was normalized to zero).
Time Frame: 2-6 weeks pre-operatively; 4-6 weeks, 6 weeks-3 months, 3-6 months, and 6-12 months post-operatively
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: meters per day
Arm/Group | Apple Watch and App
Number analyzed (Participants) | 88
meters per day
  4-6 weeks post-operatively | -792.29 (1586.98)
  3 months post-operatively: number analyzed (Participants) | 85
  3 months post-operatively | 591.27 (1502.72)
  6 months post-operatively: number analyzed (Participants) | 77
  6 months post-operatively | 915.26 (1584.86)
  12 months post-operatively: number analyzed (Participants) | 73
  12 months post-operatively | 858.99 (1705.98)

8. Primary Outcome: Patient Compliance With Wearing Apple Watch - Wear Time
Description: Average hours wear time per day across the outcome measure time frame.
Time Frame: 2-6 weeks pre-operatively
Population: Participants with available data. This outcome was evaluated on the Apple Watch and App group only (the Control group was not assigned an Apple Watch).
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Apple Watch and App
Number analyzed (Participants) | 90
hours per day | 14.05 (3.0)

9. Primary Outcome: Patient Compliance With Wearing Apple Watch - Wear Time
Description: Average hours wear time per day across the outcome measure time frame.
Time Frame: 4-6 weeks post-operatively
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Apple Watch and App
Number analyzed (Participants) | 88
hours per day | 14.26 (3.37)

10. Primary Outcome: Patient Compliance With Wearing Apple Watch - Wear Time
Description: Average hours wear time per day across the outcome measure time frame.
Time Frame: 6 weeks-3 months post-operatively
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Apple Watch and App
Number analyzed (Participants) | 85
hours per day | 14.47 (3.63)

11. Primary Outcome: Patient Compliance With Wearing Apple Watch - Wear Time
Description: Average hours wear time per day across the outcome measure time frame.
Time Frame: 3-6 months post-operatively
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Apple Watch and App
Number analyzed (Participants) | 77
hours per day | 14.49 (3.3)

12. Primary Outcome: Patient Compliance With Wearing Apple Watch - Wear Time
Description: Average hours wear time per day across the outcome measure time frame.
Time Frame: 6-12 months post-operatively
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Apple Watch and App
Number analyzed (Participants) | 73
hours per day | 14.15 (3.62)

13. Primary Outcome: Patient Satisfaction With Their Spine Care
Description: Reported as the number of participants, by response category.
Time Frame: 6 weeks post-operatively
Population: Participants who completed the survey at this time point
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Apple Watch and App
Number analyzed (Participants) | 91 | 84
Participants
  Extremely satisfied | 63 | 51
  Very satisfied | 6 | 7
  Somewhat satisfied | 20 | 23
  Neutral | 2 | 2
  Not at all satisfied | 0 | 1

14. Primary Outcome: Patient Satisfaction With Their Spine Care
Description: Reported as the number of participants, by response category.
Time Frame: 3 months post-operatively
Population: Participants who completed the survey at this time point
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Apple Watch and App
Number analyzed (Participants) | 74 | 66
Participants
  Extremely satisfied | 49 | 39
  Very satisfied | 17 | 19
  Somewhat satisfied | 4 | 4
  Neutral | 4 | 4
  Not at all satisfied | 0 | 0

15. Primary Outcome: Patient Satisfaction With Their Spine Care
Description: Reported as the number of participants, by response category.
Time Frame: 6 months post-operatively
Population: Participants who completed the survey at this time point
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Apple Watch and App
Number analyzed (Participants) | 66 | 52
Participants
  Extremely satisfied | 39 | 29
  Very satisfied | 19 | 17
  Somewhat satisfied | 5 | 2
  Neutral | 3 | 2
  Not at all satisfied | 0 | 2

16. Primary Outcome: Patient Satisfaction With Their Spine Care
Description: Reported as the number of participants, by response category.
Time Frame: 12 months post-operatively
Population: Participants who completed the survey at this time point
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Apple Watch and App
Number analyzed (Participants) | 82 | 68
Participants
  Extremely satisfied | 52 | 33
  Very satisfied | 22 | 17
  Somewhat satisfied | 4 | 13
  Neutral | 1 | 1
  Not at all satisfied | 3 | 4

ADVERSE EVENTS:
Time Frame: Up to approximately 1 year
Arm/Group | Control | Apple Watch and App
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/96
Other Adverse Events (participants affected / at risk) | 0/91 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT04379921/Prot_000.pdf
  • Statistical Analysis Plan (2025-11-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT04379921/SAP_001.pdf